CLINICAL TRIAL: NCT03162380
Title: Assessment of Occupational Stress and Well-being in French Patients Suffering From Bipolar Disorder
Brief Title: Occupational Stress and Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0138
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; occupational stress
MeSH Terms: conditions — Bipolar Disorder; Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Date collection — Date collection

SUMMARY:
Bipolar disorder is a mental disorder characterized by alternance of depressive and manic phases, separated by intercritical phases (euthymia). The majority of patients report occupation and professional difficulties. Sixty percent of bipolar patients are inactive . Indeed, according to the World Health Organisation, bipolar disorder is the second cause of days not worked.

Several factors are related to the lower professional functioning observed in bipolar patients: early age of onset, delay of diagnosis and treatment, recurrence of thymic episodes, residual symptoms and cognitive disorders during euthymia, side effects of mood stabilizers.

To our knowledge, no study has ever focused on well-being at work in French patients. However, suffering from a psychiatric disorder and the lack of support from colleagues and the hierarchy are risk factors for burnout, a growing health issue.

Patients with mental illness are often victims of stigmatization, which may involve the professional field. In addition, thymic recurrences may alter professional functioning of active patients: multiplication of work disruptions, conflicts with peers. Conversely work can be stressful, promoting thyic relapses. It is therefore essential to better understand the occupational stresses of active patients suffering from bipolar disorder in order to promote functional remission beyond clinical remission.

The aim of this study is to assess the level of stress and well-being at work in active French bipolar patients.

DETAILED DESCRIPTION:
Socio-demographic, psychiatric and occupational data of 200 bipolar patients will be collected over a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* out patients and inpatients in the Department of Emergency Psychiatry and Post Acute Care, CHU Montpellier, France
* to have completed the self-administered questionnaire on professional activity.

Exclusion Criteria:

* Deprived of liberty subject (by judicial or administrative decision)
* Protected by law (guardianship)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Bipolar disorder
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Level of occupational stress using a Likert scale | 1 day
  level of occupational stress assessed at the patient visit will be collected, from 0 (none) to 10 (maximum possible occupational stress).

SECONDARY OUTCOMES:
Presenteism during the last month using the Stanford Presenteeism Scale | 1 day
  Presenteism during the last month assessed at the patient visit will be collected
Support of colleagues and superiors using the Karasek questionnaire. | 1 day
  Support of colleagues and superiors assessed at the patient visit will be collected
Impact of work on the private sphere using the SWING scale (survey work-home interaction-Nijmegen) | 1 day
  Impact of work on the private sphere assessed at the patient visit will be collected
Balance effort - reward in using the Siegrist questionaire | 1 day
  Balance effort - reward assessed at the patient visit will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Emile OLIE, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC